CLINICAL TRIAL: NCT01890850
Title: Risk Factors Associated With Pertussis Among Infants Less Than One-year of Age
Brief Title: Study to Analyze the Risk Factors Associated With Pertussis/Whooping Cough Infection Among Infants
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Optum, Carolyn Martin and Ami Buikema (Unknown)
Responsible Party: Sponsor
Other Study IDs: 200158
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Diphtheria; Acellular Pertussis; Tetanus
Keywords: Risk factors; U.S. commercially insured population; Pertussis/whooping cough infection; Retrospective database study
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Pertussis Group: Infants less than one year of age diagnosed with pertussis/whooping cough infection within 12 months from birth (first year of life, between July 1, 2005 and September 30, 2010).
  Interventions: Other: Retrospective database study using administrative claims data
- Control Group: Infants with no evidence of pertussis/whooping cough during within 12 months from birth (first year of life, between July 1, 2005 and September 30, 2010).
  Interventions: Other: Retrospective database study using administrative claims data

INTERVENTIONS:
Other: Retrospective database study using administrative claims data — Data collection from OptumInsight proprietary research database which contains enrollment and claims data for individuals enrolled in commercial health plans.

SUMMARY:
This study aims to estimate the risk factors associated with pertussis/whopping cough infection among infants less than one year of age in a United States (U.S.) commercially insured population. The study will utilize a large research data base associated with a geographically diverse U.S. health plan not limited by one geographic area or disease outbreak to evaluate pertussis in infants between 2005 and 2010. Healthcare costs and utilization among infants with a reported diagnosis of pertussis/whooping cough stratified by the number of DTaP vaccinations received prior to infection will also be reported.

DETAILED DESCRIPTION:
This study will utilize the OptumInsight proprietary research database which contains enrollment and claims data for individuals enrolled in commercial health plans to estimate the measureable demographic, clinical and historical economic risk factors that may be associated with medically diagnosed pertussis/whooping cough infection among commercially insured infants less than one-year of age. Healthcare costs and utilization among infants with a reported diagnosis of pertussis/whooping cough will be stratified by the number of DTaP vaccinations received prior to infection.

ELIGIBILITY:
Inclusion Criteria:

* Date of birth between July 1, 2005 and September 30, 2010.
* Enrollment in a commercial health plan within one month of birth.
* Known sex and geographic region.
* Infants will be included as a pertussis/whooping cough case if they meet the diagnosis criteria Infants not identified as a pertussis/whooping cough case are eligible for inclusion as a control.

Exclusion Criteria:

• Enrollment does not include medical and pharmacy coverage.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants less than one-year of age born between 2005 and 2010 in a U.S. commercially insured population contained within the optum propertity database
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Assessment of claim identified pertussis/whooping cough | Up to one year
  The endpoint(s) for the primary objective are the odds ratios associated with factors modelled in a logistic regression (conditional logit model) where the outcome is the diagnosis of pertussis/whooping cough. Demographic, economic and clinical risk factors available in the administrative claims database and potentially associated with pertussis/whooping cough infection will be estimated. Covariates will be determined based on clinical rationale and statistical significance.
Assessment of health care resource utilization | Up to one year
  Health care resource utilization (e.g. ambulatory visits, emergency department visits, inpatient hospitalizations, length of stay) will be calculated for infants with a reported diagnosis of pertussis/whooping cough stratified by the number of DTaP vaccinations received prior to infection.
Assessment of health care costs | Up to one year
  Health care costs will be computed as the combined health plan and patient paid amounts in the post-index period. Costs will be calculated as a total costs, medical costs, pharmacy costs, ambulatory costs, emergency costs and other costs and split by those occurring prior to the index date and those in the follow-up period. Costs will be adjusted to 2012 U.S. dollar values using the Medical Care Consumer Price Index.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Masseria C, Martin CK, Krishnarajah G, Becker LK, Buikema A, Tan TQ. Incidence and Burden of Pertussis Among Infants Less Than 1 Year of Age. Pediatr Infect Dis J. 2017 Mar;36(3):e54-e61. doi: 10.1097/INF.0000000000001440. PMID 27902648